CLINICAL TRIAL: NCT07152730
Title: An Open-label Trial Investigating the PK of Gonadotropin Releasing Hormone (GnRH) Administrated Subcutaneously Via the OmniPod Delivery System in Healthy Female Subjects
Brief Title: A Study to Measure Pharmacokinetic (PK) Concentrations of Gonadotropin-Releasing Hormone Delivered by the OmniPod Pump
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate development activities was based on business needs and unrelated to any safety or efficacy concerns.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000438; U1111-1313-1848 (Other: WHO)
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Amenorrhea; Fertility; Infertility
Keywords: Amenorrhea; Lutrepulse; Fertility; OmniPod
MeSH Terms: conditions — Amenorrhea; Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (single dose) (Experimental): Single-dose (1 pulse) LUTREPULSE Omnipod 20ug/pulse
  Interventions: Drug: Lutrepulse
- Group B (multiple doses) (Experimental): Part 1 - Single dose (1 pulse) LUTREPULSE Omnipod 20ug/pulse Part 2 - multiple doses (6 pulse) LUTREPULSE Omnipod 20ug/pulse
  Interventions: Drug: Lutrepulse

INTERVENTIONS:
Drug: Lutrepulse — Lutrepulse administered via the OmniPod delivery pump

SUMMARY:
One of the Causes of Amenorrhea is hypothalamic amenorrhea, which is a deficiency in the amplitude and/or frequency of endogenous Gonadotropin-releasing hormone (GnRH) Pulses. The results of this leads to anovulation and cessation of the menstrual cycle. Pulsatile GnRH has been widely used in the United States (US), Canada, and Europe for almost 40 years in the treatment of primary hypothalamic amenorrhea. It has a favorable safety profile and a high degree of effectiveness in enabling ovulation and spontaneous pregnancy. At the moment there are no other GnRH products on the market, nor are there any other drugs marketed for induction of ovulation in women with primary hypothalamic amenorrhea in the US, creating a clear unmet medical need. The goal of this trial is to characterize the exposure variability of GnRH when administered via the OmniPod.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects 18 to 40 years old (both included).
2. Body mass index (BMI) between 18 and 30 kg/m2 (both included).
3. Regular menstrual cycles of 24 to 35 days (both included).

Exclusion Criteria

1. Any medical condition, which in the judgment of the investigator, may interfere with the absorption, distribution, metabolism, or excretion of gonadotropin-releasing hormone (GnRH).
2. Use of any hormonal contraceptives, growth hormone, insulin or thyroid hormone replacement therapy 30 days prior to dosing in this trial.
3. Previously known or suspected hypersensitivity to GnRH.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Cmax: maximum observed plasma concentration from Part 1- Pulse 1 | Up to 5 days
AUC0-t: area under the concentration-time profile to the last quantified concentration from Part 1- Pulse 1 | Up to 5 days
AUC0-infinity: area under the concentration-time curve to infinity from Part 1- Pulse 1 | Up to 5 days

SECONDARY OUTCOMES:
tmax: time to maximum plasma concentration from Part 1- Pulse 1 | Up to 5 days
λz; terminal elimination rate constant from Part 1- Pulse 1 | Up to 5 days
t½; terminal elimination half-life from Part 1- Pulse 1 | Up to 5 days
Cmax: maximum observed plasma concentration from Part 2 - Pulse 6 | Up to 4 days
AUC0-t: area under the concentration-time profile to the last quantified concentration from Part 2 - Pulse 6 | Up to 4 days
AUCtau: area under the concentration-time profile at steady-state from Part 2 - Pulse 6 | Up to 4 days
tmax: time to maximum plasma concentration from Part 2 - Pulse 6 | Up to 4 days
λz; terminal elimination rate constant from Part 2 - Pulse 6 | Up to 4 days
t½; terminal elimination half-life from Part 2 - Pulse 6 | Up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ferring Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No